CLINICAL TRIAL: NCT06207708
Title: Role of Baseline Sarcopenia in Determining Acute Toxicity for Head and Neck Cancer Patients Treated with Curative Hadrontherapy: a Prospective Monoinstitutional Study
Brief Title: Sarcopenia in Head and Neck Cancer Patients Treated with Curative Hadrontherapy
Status: Completed | Type: Observational
Sponsor: CNAO National Center of Oncological Hadrontherapy (Other)
Responsible Party: Sponsor
Other Study IDs: CNAO 56 2023
Record Dates: First submitted 2024-01-03; First posted 2024-01-17 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Head and Neck Cancer
Keywords: particle therapy; head neck cancer; sarcopenia; hadrontherapy
MeSH Terms: conditions — Head and Neck Neoplasms; Sarcopenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: questionnaires QLQ-FA12, Mini Nutritional Assessment Short Form, Nutritional Risk Screening, diet questionnaire of frequency, ,body mass index measurement — the patient is administered with questionnaires focused on diet, fatigue, nutrition screening and on body mass index at the beginning and at the end pf particle therapy radiation treatment
Diagnostic Test: blood biomarkers — as per clinical routine, hemoglobin, lymphocytes, albumin and NLR will be collected

SUMMARY:
The study focuses on the impact of sarcopenia on acute and late toxicities in head and neck tumor affected patients treated with particle therapy.

DETAILED DESCRIPTION:
To evaluate in HNC patients treated with particle therapy the impact of SP (measured by low skeletal muscle mass at the C3 vertebral body) on toxicity profile assessed according to NCI's Common Terminology Criteria for Adverse Events CTCAE (version 5.0), defined as:

* Acute toxicity: within 3 months from the beginning of particle RT
* Late toxicity: more than 6 months after the end of particle RT. To investigate possible association between SP and nutritional

ELIGIBILITY:
Inclusion Criteria:

* All HNC histologies and stages
* Histological and/or radiological diagnosis of head and neck tumors
* The patient is able to give consent
* Definitive/postoperative treatment with curative intent
* Age >18 years
* KPS> 80

Exclusion Criteria:

* Plurimetastiatic disease
* Palliative intent and re-irradiation treatments
* Known cases of any psychiatric and neurological diseases leading to disability (eg, manic disorder, schizophrenia etc..), which could impair compilation of questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A sample of 70 patients of which 40% showing baseline sarcopenia will be recruited. The population is composed by head and neck patients treated with particle therapy, both carbon ions and protons.
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2023-04-18 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
skeletal muscle strength mass (SMM) | before starting hadrontherapy treatment
  measurement of sarcopenia to evaluate the development of the affection

CONTACTS AND LOCATIONS:
Overall Officials: Rossana Ingargiola, MD, Principal Investigator — CNAO National Center of Oncological Hadrontherapy
Locations (1):
- CNAO, Pavia, Pv, Italy

IPD SHARING:
Plan to Share IPD: No